CLINICAL TRIAL: NCT02349854
Title: Neurobiology of the Scalp in Seborrheic Dermatitis
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Sponsor
Other Study IDs: H-31892
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Seborrheic Dermatitis
Keywords: pruritus; itch; skin; scalp; seborrheic dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic; Pruritus | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Scalp biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: patients with scalp itch and seborrheic dermatitis who will get biopsy
  Interventions: Procedure: Biopsy
- Controls: patients without scalp itch and without seborrheic dermatitis who will get biopsy
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — 1 scalp biopsy will be done at the site of central sensitization testing, according to standard of care practices. First, the site will be anesthetized and within this area, 2 immediately adjacent (ie contiguous) punch biopsies will be taken-2mm & 3mm. Both will be closed simultaneously using either (i) non fast-absorbing gut sutures, requiring a 10-14 day follow-up visit for suture removal; (ii) fast absorbing gut sutures that will not require a subsequent suture removal visit, or (iii) gel foam without stitches that also does not require a suture removal visit. Wound care instruction will be discussed with patient. The patient will be instructed to apply petroleum jelly at least 3 times per day to the biopsy site, reflecting standard of care clinical care at BMC.

SUMMARY:
Seborrheic dermatitis is a common, inflammatory skin condition that causes flaky, white to yellowish scales to form on oily areas such as the scalp or inside the ear. These scales can occur with or without underlying reddened skin. In addition to causing psychological distress, low self esteem, and embarrassment, seborrheic dermatitis is associated with scalp pruritus (itch). Treatment modalities exist to control scalp flaking and itch associated with seborrheic dermatitis, although such therapies often lose efficacy over time. As seborrheic dermatitis is a chronic (life-long) condition, better treatments are needed. The investigators propose to better characterize in subjects with seborrheic dermatitis involving the scalp versus normal scalp controls: (a) the clinical characteristics of the associated itch and (b) the pattern of nerve innervation to the scalp. In this way, the investigators hope to get a comprehensive understanding of the factors causing scalp itch with the aim that this information will create new candidates to which treatment modalities can be designed. At least 12 (up to 20) subjects and similar number of control subjects without disease will have one clinic visit including questionnaires, testing of sensation on the scalp, and biopsy of the scalp.

DETAILED DESCRIPTION:
Seborrheic dermatitis (SD) is a common skin disorder that mainly affects the scalp, causing scale, itch, and red skin. Dandruff, a subset of SD, shows scale and itch in the absence of associated red skin. Seborrheic dermatitis can occur on many different body areas, including the scalp, eyebrows, eyelids, creases of the nose, lips, behind the ears, in the outer ear, and middle of the chest. On the scalp, SD is commonly associated with pruritus (itch). Multifactorial theories have been proposed regarding the pathogenesis of SD, and these include irritation from a skin-based yeast called malessizia, overproduction of sebum by sebaceous glands in the affected skin areas, and individual variability. Specifically, malassezia produce free fatty acids from sebaceous gland-produced triglycerides, and these free fatty acids have an "irritant" (ie, non-immunologic) effect in those patients with a "susceptible predisposition." Other factors associated with flares of SD include stress, fatigue, weather extremes, infrequent shampoos or skin cleaning, use of lotions that contain alcohol, skin disorders (such as acne), obesity, neurologic conditions (including Parkinson's disease, stroke, and head injury), and HIV infection. What role, if any, such factors play in the etiology of scalp pruritus in patients with SD is not known. Furthermore, itch is signaled by specific subsets of nerves in the skin and whether pruritus of SD results from alteration of these nerves by the underlying inflammatory state is unknown. Moreover, pruritus from the skin can be a result of peripheral sensitization, where skin-derived signals activate nerves in the skin to send increased nerve signals into the central nervous system. Pruritus sensed in the skin can also be a result of altered central-nervous system processing of skin-derived nerve signals, such as when skin-derived touch or pain is misperceived as itch by the central nervous system. Whether itch in patients with SD is a result of peripheral and/or central sensitization is also not unknown. Understanding this distinction has therapeutic implications, in that itch that is a result of misprocessing by the central nervous system will not be adequately treated, in the short term, by skin-administered topical therapies.

To better understand the etiology of scalp pruritus in subjects with SD, we will determine the clinical characteristics of scalp pruritus in subjects with SD compared with normal controls, as well as to determine the relationship between scalp pruritus and changes in cutaneous innervation.

METHODS:

This exploratory and pilot study has only a single planned visit to the outpatient Dermatology clinic in Shapiro center.

Subjects who carry the diagnosis of seborrheic dermatitis and scalp itch, or controls who don't, (either internally referred through routine visits to outpatient Dermatology clinics at BMC or externally referred from outside providers or who respond to recruitment techniques) will undergo an initial phone screening to review inclusion and exclusion criteria. This screening will involve anonymous screening questions without collection of personal health information. Subjects/controls that meet the criteria to be eligible for the study will then be asked if they are willing to come to BMC for the single study visit. Those subjects/controls that then agree to be scheduled will next be told that we are seeking informed consent by phone for the following minimal risk procedures in preparation for the study visit:

1. to place a unique patient code identifier on the screening form and
2. if they are willing to stop using any topical scalp treatments for seborrheic dermatitis/dandruff as well as (c) to stop any prn or elective use of prescribed or over-the counter antihistamines for at least 3 weeks before their scheduled visit.

(d) if they are willing not to wash their hair for at least 48 hours prior to the visit.

The consent process will include highlighting that the individual can stop the "washout" at anytime. Those subjects/controls, after undergoing informed consent process read to them over the phone, that agree to (a) and (b) and (c) above, will then be scheduled for a one hour visit at the outpatient Dermatology floor during a non-clinic time.

At this visit, all subjects/controls will first undergo the following:

1. Visual and non-invasive inspection of the scalp
2. Completion by the patient of a visual analogue scale (VAS) score to measure degree of scalp pruritus over the past week. This VAS form will have no identifiable health information.
3. Review of the inclusion/exclusion criteria answers they provided over the phone, that after informed consent by phone at the time they gave those answers, they agreed to allow us to store with a unique subject/control identifying code.

The above 3 minimal risk procedures (one of which the patients have already provided informed consent for), will happen before "study visit screening" (described in detail in Screening Section 20.0 below) and the second informed consent process is performed. This order is to respect the patient's time. If they no longer meet inclusion/exclusion criteria based on the above minimal risk screening, they will not be eligible for the study and so would then have unnecessarily undergone additional screening as well as an informed consent process.

After obtaining written informed consent to participate in the study, the following will occur:

1. Female subjects of child-bearing potential will take a urine pregnancy test.
2. Subjects/controls will fill-out a questionnaire for pruritus and a questionnaire that contains additional targeted questions related to their scalp itch and hair care practices
3. Investigators will assess scalp to identify involved, pruritic sites along EEG lead axis T3-O1 or, secondarily, along EEG lead axis C3 to Pz. EEG testing is a standard non-invasive neurologic test in which scalp electrodes are placed in well-defined and specified positions on the scalp. We will not be doing an EEG or using electrodes. We are simply using the anatomic landmarks specified for EEG placement to allow uniform selection of scalp areas to test and biopsy.
4. Digital photographs of the patient's head, focusing on the scalp will be taken.
5. At the selected scalp site, an investigator will perform the following tests for central sensitization, at the selected scalp site (see below for methods for these tests):

   * Warm heat (methods section below explains this procedure) to assess it is or is not felt as itch using 3 mm diameter metal probe
   * Alloknesis (brush to itch: if possible on scalp with hair)
   * Hyperknesis (enhanced sensation of itch to pinprick)
   * Duration of itch elicited by insertion of a cowhage spicule into the scalp (if possible on scalp with hair). This procedure is described in detail below.
6. The investigator will then perform a single scalp biopsy procedure at the site of central sensitization testing, according to standard of care practices. The 2mm specimen will be placed into formalin for routine paraffin-embedding. The 3mm specimen will be placed into a special fixative that optimizes immunohistochemistry on frozen sections to detect antigens expressed by nerves. These specimens will be labeled with the subjects/control's unique identifying code only and without personal health information.

This one visit completes the subjects/control's entire participation in the study. No additional visits will be scheduled (unless the individual has opted for suture option and removal of these sutures at BMC) but the subject/control will be provided the contact information of the investigator in the rare event that the subject/control requires further care as a complication of the biopsy procedure, such as bleeding, persistent pain, infection, and/or failure to heal.

In all biopsies, the density and distribution of different subsets of cutaneous nerve fibers will be determined by immunohistochemistry in the frozen-fixed tissue and the presence or absence of histopathologic features of seborrheic dermatitis will be evaluated in the paraffin-embedded tissue. Left over tissue from either the frozen and/or the paraffin-embedded tissue will be saved in a repository if the individual consents, and the storage of these tissues and safeguards are described in detail in the tissue banking section of the BMC approved IRB protocol.

Estimated Duration of Enrollment (how long will it take to recruit the required sample size): One year.

Estimated Duration of Entire Study (estimated duration from initial IRB approval through data analysis to close of study): Two years Sample Size- Total=60 patients with scalp itch and seborrheic dermatitis =30

* consent and/or fully participate in study = 20
* expected drop outs withdrawal and terminations = 5
* screened and not enrolled = 5 patients without scalp itch and without seborrheic dermatitis =30
* consent and/or fully participate in study = 20
* expected drop outs withdrawal and terminations = 5
* screened and not enrolled = 5

Sample Size Justification:

Although the proposed study is exploratory in intent and does not require a formal power statement, we can nonetheless estimate power for the primary outcome of no central sensitization in patients with seborrheic dermatitis versus controls for the planned sample size of 20 subjects. The expected average mean score for a patient with central sensitization is 3 out of 10 and for a control patient 1 out of 10 with a standard deviation of 1. Therefore, for there to be no difference between both groups, we would expect both groups to have a mean score of 1 with a standard deviation of 1. In this case, if there is truly no difference between the control and experimental group (ie, no central sensitization), then 36 total patients (18 per group) are required to be 80% sure, 40 total patients (20 per group) are required to be 85% sure, and 44 total patients (22 per group) are required to be 90% sure, that the 90% two-sided confidence interval will exclude a difference in means of more than 1. We feel that in this instance, certainty over 80% will be clinically meaningful and have opted for 40 instead of 36 to better ensure the date achieves at least 80% certainty.

For the total number per cohort, some number of patients will contact us and undergo anonymous screening questions without collection of personal health information. This number is difficult to predict, and those patients that do not meet eligibility criteria based on the answers to these anonymous screening questions, are not included in either cohort as there is no risk to them, again because no personal health information is being collected.

Data Analysis:

The proposed study design is one in which for each one of the three specific aims described above, there is one dependent variable (outcome) and 1 independent variable (2 independent populations: subjects with seborrheic dermatitis and scalp itch and controls without scalp itch or seborrheic dermatitis). For non-normal data, we intend to use a non-parametric test, such as the Mann Whitney or Wilcoxon rank sum test to assess for statistical differences between the medians between these populations. In addition, we will use non-parametric analysis, such as the Spearman correlation to correlate results of the skin testing with results of the immunohistochemical counts of nerves. If in fact distributional assumptions are met to allow parameteric analysis, we will use a 2 independent sample t-test to assess for statistical differences between the means.

ELIGIBILITY:
Inclusion Criteria:

Study Subjects

* Individuals 18 years or older
* Pruritus measured by VAS score for scalp itch greater than or equal to 30 in past week and "dandruff" without skin changes or erythema but with histologic evidence of at least focal or mild epidermal spongiosis
* Pruritus measured by VAS score for scalp itch greater than or equal to 30 in past week and seborrheic dermatitis, including histologic evidence of at least focal or mild epidermal spongiosis
* No topical anti-pruritic treatments and no prescribed or over-the-counter topical seborrheic dermatitis treatments for at least 3 weeks before initiation of study, including antifungal shampoos, tar or urea-containing shampoos, selenium sulfide or zinc-containing shampoos, or topical steroids
* Willingness to forgo elective (ie PRN) use of systemic over-the-counter or prescribed antihistamines to treat conditions other than chronic pruritic skin diseases (for example, seasonal allergies) for at least 3 weeks before initiation of the study

Control Subjects

* Individuals 18 years or older
* No pruritus of the scalp as measured by VAS score for scalp itch less than 30 in past week and no "dandruff" or scalp skin changes or erythema and no histologic evidence of at least focal or mild epidermal spongiosis
* No pruritus of the scalp as measured by VAS score for scalp itch less than 30 in past week and no seborrheic dermatitis, including no histologic evidence of at least focal or mild epidermal spongiosis
* No topical anti-pruritic treatments and no prescribed or over-the-counter topical seborrheic dermatitis treatments for at least 3 weeks before initiation of study, including antifungal shampoos, tar or urea-containing shampoos, selenium sulfide or zinc-containing shampoos, or topical steroids
* Willingness to forgo elective (ie PRN) use of systemic over-the-counter or prescribed antihistamines to treat conditions other than chronic pruritic skin diseases (for example, seasonal allergies) for at least 3 weeks before initiation of the study

Exclusion Criteria:

* Individuals with the diagnosis of psoriasis or evidence of psoriasis in other non-scalp body areas
* Individuals with evidence of any primary scarring alopecia (active or inactive).
* Individuals with non-dermatologic scalp itch, including scalp itch with no scale (ie dandruff) or erythema, individuals with senile pruritus of the scalp, or scalp dysthesias (such as in the setting of anxiety/mood disorders).
* Individuals on anti-depressant medication specifically to treat pruritus. (Patients on anti-depressants for non-pruritus reasons and that meet the VAS criteria for itch will be included).
* Individuals with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Individuals unable to read and/or comprehend the questionnaires utilized in this study
* Individuals that present with haircare practices associated with scarring alopecias, such as but not limited to, hot combing, chemical relaxers/straighteners, and tight braiding
* Individuals with an allergy and/or history of adverse reaction to lidocaine used for the scalp biopsy
* Any use of systemic anti-pruritic or anti-fungal treatments in the 3 weeks prior to initiation of the study, including systemic corticosteroids, immunosuppressive agents, phototherapy, or antihistamines (in the setting of chronic use for anti-pruritic therapy, such as chronic urticaria)
* Women who are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dermatology clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percentage of vasodilatory peptidergic nerve fibers in the papillary dermis versus total nerves in the papillary dermis in control versus diseased scalp | one year
  Hypothesis: Scalp pruritus in patients with seborrheic dermatitis is associated with a change in the neuropeptide identity of nerves at the dermal-epidermal junction (DEJ).

SECONDARY OUTCOMES:
Presence or absence of brush-stoke induced pruritus in disease versus control skin | one year
  (i) assessment of brush-stroke induced pruritus: involved and non-involved skin areas chosen for other tests of central sensitization will be stroked smoothly and lightly by a cotton swab or a small paint brush at a rate of 1 Hz. The participants will be asked to report the evoked sensation.
Duration (minutes) of cowhage-spicule induced pruritus in diseases versus control skin | 1 year
  Pinprick stimuli will be applied to the scalp skin with a series of probes: 2 mL syringe barrel containing a free-floating sterile 27-gauge cannula above which is 1 of these weights: 1.0, 2.3, 3.7, 8.6, or 14.8 g. Each probe will be laid down gently on the skin to prevent damage, and then held for 2 seconds. The subjects will be asked to describe the quality and intensity of the evoked sensation. The intensities of itch and pain will be reported separately on a numeric scale ranging from 0 (no sensation) to 10 (maximal sensation imaginable). This mode of application was reported in a previously published study in patients with atopic dermatitis (Ikoma et al, 2004. Neurology; 62: 212-7)to produce maximal itch sensation of less than 3 and maximal pain sensation of less than 4 on a numeric scale ranging from 0 (no sensation) to 10 (maximal sensation imaginable). This procedure will be repeated 10 times with each load in the area of the scalp that will be selected for skin biopsy.
Amount of pin-pressure induced pruritus in diseased versus control skin | one year
  Pinprick stimuli will be applied to the scalp skin with a series of probes: 2 mL syringe barrel containing a free-floating sterile 27-gauge cannula above which is 1 of these weights: 1.0, 2.3, 3.7, 8.6, or 14.8 g. Each probe will be laid down gently on the skin to prevent damage, and then held for 2 seconds. The subjects will be asked to describe the quality and intensity of the evoked sensation. The intensities of itch and pain will be reported separately on a numeric scale ranging from 0 (no sensation) to 10 (maximal sensation imaginable). This mode of application was reported in a previously published study in patients with atopic dermatitis (Ikoma et al, 2004. Neurology; 62: 212-7)to produce maximal itch sensation of less than 3 and maximal pain sensation of less than 4 on a numeric scale ranging from 0 (no sensation) to 10 (maximal sensation imaginable). This procedure will be repeated 10 times with each load in the area of the scalp that will be selected for skin biopsy.
Amount of thermal (sensation of mildly painful and non-damaging heat)-induced itch in diseased versus control skin | one year
  Thin metal rod (diameter, ~2-3 mm) will be preheated to 41, 46, or 49 °C in a temperature-controlled water bath and then sequentially applied perpendicularly to the skin and held for 10 seconds. These temperatures with this short length of application are not enough to cause thermal damage to the skin. The maximal reported sensation was 3.5 for pain and 2.5 for itch on the above 0-10 scale. The subjects will be asked to rate the intensities of the evoked itch and pain every 2 secs from 0 (first placement) to 20 sec after placement. This procedure will be performed once in the area of the scalp that will be selected for skin biopsy. The area under the curves for both itch and pain perception plotted against time will be compared for each site tested.
Percent of autonomic nerves to total nerves innervating adnexal structures in diseased versus control skin | one year
  Hypothesis: Scalp pruritus in patients with seborrheic dermatitis is associated with a change in the distribution or number of autonomic nerves innervating adnexal structures.

CONTACTS AND LOCATIONS:
Overall Officials: Deon Wolpowitz, MDPhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No